CLINICAL TRIAL: NCT01399476
Title: Endoscopic Submucosal Tunnel Dissection for Endoluminal Partial Myotomy of the Lower Esophageal Sphincter for Achalasia
Brief Title: Endoscopic Myotomy of the Lower Esophageal Sphincter for Achalasia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Lee Swanstrom, Lee Swanstrom, MD, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1056
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Achalasia
Keywords: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic Myotomy (Experimental)
  Interventions: Procedure: Endoscopic Myotomy; Procedure: Endoscopic Myotomy for treatment of achalasia

INTERVENTIONS:
Procedure: Endoscopic Myotomy — Patients will receive the surgical procedure described in the summary (POEM).
  Other Names: POEM
Procedure: Endoscopic Myotomy for treatment of achalasia — Surgical procedure
  Other Names: POEM

SUMMARY:
This is a study of the safety and efficacy of a new surgical procedure using endoscopic instruments and a tunneling technique to reach the LES for dissection. We hypothesize that this technique provides an incisionless, less invasive option with similar functional outcome compared to standard Heller myotomy.

DETAILED DESCRIPTION:
By the endoscopic creation of an esophageal submucosal tunnel the inner circular muscle layer can be easily visualized. In contrast to conventional Heller myotomy, the dissection of only the inner circular esophageal muscle layer leaves the outer longitudinal muscle layer intact. Thereby, post-interventional reflux disease should be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo general anesthesia
* Age > 18 yrs. of age and < 85 yrs. of age
* Ability to give informed consent
* Candidate for elective Heller myotomy

Exclusion Criteria:

* Previous mediastinal or esophageal surgery
* Contraindications for esophagogastroduodenoscopy
* BMI > 45

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Improved quality of life as defined by survey pre and post surgery | six months
  patients diagnosed with achalasia will be given a quality of life survey before surgery and again six months after surgery.

SECONDARY OUTCOMES:
Negative pH test | six months
  Patients will be required to have 24 hour pH testing after surgery.
Bleeding | 1 year
  recorded blood loss will be taken during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lee L Swanstrom, MD, Principal Investigator — The Oregon Clinic
Locations (1):
- The Oregon Clinic, Portland, Oregon, United States

REFERENCES:
- [Derived] Kurian AA, Dunst CM, Sharata A, Bhayani NH, Reavis KM, Swanstrom LL. Peroral endoscopic esophageal myotomy: defining the learning curve. Gastrointest Endosc. 2013 May;77(5):719-25. doi: 10.1016/j.gie.2012.12.006. Epub 2013 Feb 5. PMID 23394838